CLINICAL TRIAL: NCT03530384
Title: Training Inhibition in Alcohol Use Disorder: an add-on Randomized Controlled Trial
Brief Title: Training Inhibition in Alcohol Use Disorder
Acronym: TRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P160930J; 2017-A03558-45 (Other: ANSM)
Record Dates: First submitted 2018-04-13; First posted 2018-05-21 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-03

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training (Experimental): Computerized cognitive training program targeting inhibitory control
  Interventions: Other: Cognitive training
- Control Training (Sham Comparator): A sensorial program with similar conditions, but targeting visual acuity, considered as neutral in the addiction field
  Interventions: Other: Control training

INTERVENTIONS:
Other: Cognitive training — Computerized cognitive training targeting inhibitory control of motor response used during 45 minutes sessions twice a week for 6 weeks
  Arms: Cognitive training
Other: Control training — Fictitious computerized training used during 45 minutes sessions twice a week for 6 weeks
  Arms: Control Training

SUMMARY:
More and more studies aim to improve neurocognitive functioning in alcohol use disorder, but very few studies have focused on training-inhibitory-control efficacy on alcohol intake. Our program relies on a comprehensive model of addiction considering inhibition deficit as the hallmark of addiction. Our program proposes inhibition training on a task which does not refer to alcohol, combined with a debriefing promoting transferability of the enhanced skill and psychoeducation. In this perspective of aiming to retrain deficits involved in addiction in itself and not only due to alcohol toxicity. We propose an add-on single-blinded randomized controlled trial, in alcohol use disorder, assessing the efficacy of a computerized cognitive training program targeting inhibition as compared to treatment as usual.

DETAILED DESCRIPTION:
Our hypothesis is that a computerized program aiming to retrain deficits involved in addiction in itself and not only due to alcohol toxicity i.e.inhibition training on tasks which do not refer to alcohol, combined with a debriefing promoting transferability of the enhanced skills, in addition to treatment as usual, is more effective than a control condition in addition to treatment as usual.

The program is a computerized cognitive training targeting inhibitory control of motor response (Scientific Brain Training®). The tasks included in the program have been selected and modified to target inhibition processes. The tasks are "find your way", "Don't fall in the trap", "Under pressure", "gulf-stream", "catch the ladybird" and an additional task: "Color and word Stroop test".

The program must be dispensed twice a week with at least in the week one session on site, the other either on site or at home via an application to download, during 6 weeks.

The duration for one session is 45 minutes, including:

* 30 minutes performing the selected modules with increasing level of difficulty corresponding to their personal improvement. The patient will be able to choose within the selected modules the ones they want to perform during one session.
* 15 minutes of group (for onsite sessions) debriefing mediated by a neuropsychologist. The debriefing will follow a semi-structured framework including a focus on the emotion associated with the task completion and a focus on the transferability of the tasks in the patient real life.

Control condition: A sensorial program with similar conditions (45 minutes sessions twice a week), but targeting visual acuity, considered as neutral in the addiction field.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65;
* With a current alcohol use disorder, according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5), and with at least a high drinking risk level (men: alcohol consumption >60 g/day; women >40 g/day), in the last 4-week drinking period ;
* Who must be abstinent since 7 to 30 days at the inclusion visit, no matter their drinking goal for the following period ;
* Who should not have been administered benzodiazepines since at least 3 days at the inclusion visit (to avoid interference with alcohol intoxication or withdrawal medication on the neuropsychological assessments in one hand, and any recall bias on drinking ones in the other hand);
* Affiliated to social security;
* Who has given a written informed consent.

Exclusion Criteria:

Will not be included patients:

* With current alcohol withdrawal symptoms (Cushman score > 3) at the inclusion visit;
* With dual addiction (excluding tobacco);
* With psychiatric comorbidity (psychotic disorders, current manic/hypomanic episode, current major depressive episode), as assessed with the Mini International Neuropsychiatric Interview (MINI), Alzheimer disease, Korsakoff syndrome, mental retardation, or any condition that may significantly alter the computerized-task completion, as assessed by the clinician's judgment;
* Unable or unwilling to comply with the protocol requirements and/or unwilling to sign an informed consent form.
* Deprived of liberty or under legal protection measure.
* Pregnant or lactating woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
The reduction in number of heavy drinking days between the last drinking 4-week period and 6 weeks, assessed with the Time Line Follow Back (TLFB). | 6 weeks
  The number of heavy drinking days (HDD) is defined as a day with an alcohol consumption ≥60 g for men and ≥40 g for women.

SECONDARY OUTCOMES:
Change in total alcohol consumption (g/day) between T1 and - T2, -T3 assessed with the TLFB | 12 weeks
Change in number of heavy drinking days between T1 and -T3 assessed with the TLFB | 12 weeks
Change in Alcohol Quality of life scale between T1 and -T2, -T3 | 12 weeks
Change in Clinical Global Impression scale (CGI) severity between T1 and -T2, -T3 | 12 weeks
Change in Difficulties in Emotion Regulation Scale-Impulse (DERS-IMPULSE ) between T1 and -T2, -T3 | 12 weeks
Change in Stop Signal Reaction Time (SSRT) between T1 and -T2, T3 | 12 weeks
Change in Stop-signal delay (SSD) from the Stop Signal Task (SST) between T1 and -T2, T3 | 12 weeks
Change in Wechsler Adult Intelligence Scale (WAIS) between T1 and -T2, -T3 | 12 weeks
Change in Corsi test between T1 and -T2, -T3 | 12 weeks
Change in Brixton test between T1 and -T2, -T3 | 12 weeks
Change in Trail Making Test (TMT) between T1 and -T2, -T3 | 12 weeks
Change in Verbal fluencies test between T1 and -T2, -T3 | 12 weeks
Description of the influence of catechol-O-methyltransferase (COMT) variant on efficacy | one day
  Genotyping of catechol-O-methyltransferase (COMT)

CONTACTS AND LOCATIONS:
Locations (1):
- Paul Brousse Hospital, Villejuif, France